CLINICAL TRIAL: NCT06133933
Title: Total Shoulder Arthroplasty Preoperative Pain Threshold Prospective
Brief Title: Total Shoulder Arthroplasty Preoperative Pain Threshold and Association With Postoperative Opioid Consumption
Status: Enrolling by invitation | Type: Observational
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Catherine Fedorka MD, Orthopaedic Surgeon, Assistant Professor of Orthopaedic Surgery, Assistant Program Director, Orthopaedic Surgery Residency Program, The Cooper Health System
Other Study IDs: IRB 21-087
Record Dates: First submitted 2023-07-26; First posted 2023-11-18 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Total Shoulder Arthroplasty; Postoperative Pain; Opioid Use
Keywords: Total Shoulder Arthroplasty; Postoperative Pain; Postoperative Satisfaction; Opioid consumption
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Patients will have their preoperative pain threshold measured and complete postoperative pain journal, pill count, VAS, SF-12, SANE, and Satisfaction Survey in addition to the routine standard of care following perioperative management of total shoulder arthroplasty patients.
  Interventions: Device: Pain Threshold using algometer/dolorimeter

INTERVENTIONS:
Device: Pain Threshold using algometer/dolorimeter — These patients who consent to participation in the study will receive a preoperative pain threshold measured using a pain algometer/dolorimeter. We will rely on the completion of the questionnaires, opioid consumption journal, and surveys to establish a correlation between pre-operative pain threshold and post-operative outcomes.

SUMMARY:
The purpose of this prospective research study is to evaluate the effects of preoperative pain threshold using a pressure algometer and its effects on postoperative patient satisfaction, return to work, and opioid consumption following Total Shoulder Arthroplasty (TSA). Participants will have their pain threshold measured at the preoperative visit. Postoperatively, they will be followed for 3 months and complete a pain journal for 2 weeks, record their medications consumed, and complete surveys at 2 weeks, 6 weeks, and 3 months. The study team will rely on the completion of the questionnaires, opioid consumption journal, and surveys to establish a correlation between pre-operative pain threshold and post-operative outcome.

DETAILED DESCRIPTION:
Prior to undergoing total shoulder arthroplasty (TSA), it is important to counsel the patient on what the postoperative period will look like. Important factors that patients must consider include recovery time, amount of experienced pain, and risks for complications. A lower preoperative pain level has been shown to be a strong predictor of less postoperative pain, less opioid consumption, and greater patient satisfaction. However, pain is relative and typically quantified on a scale of 1-10. The pressure pain algometer is a tool that allows for the quantification of pain threshold and has demonstrated strong reliability with low inter-observer error. The pressure pain algometer has been used to determine preoperative pain thresholds in previous human studies and has been regarded as a suitable tool for assessing pain. Despite the use of this technique in the current literature, data on the application of this tool in Total Shoulder Arthroplasty (TSA) is lacking. There is no current study that has studied the use of preoperative pain thresholds using a pressure pain algometer and its correlation of patient satisfaction, and opioid consumption in TSA patients. This study will be important in closing the knowledge gap in the current literature and provide a better understanding of the usefulness of assessing preoperative pain thresholds with a pressure pain algometer on determining postoperative patient satisfaction, and opioid consumption in patients undergoing total shoulder arthroplasty.

This is a prospective, non-randomized observational study. There will only be one group, the treatment group, consisting of patients undergoing Total Shoulder Arthroplasty (TSA). The study team will recruit patients using a screen for patients who meet inclusion criteria in the institutional electronic medical record platform, EPIC, or recruit patients via physician referral. Inclusion criteria include all patients over 18 years of age who are undergoing TSA. When an eligible patient is selected, the study team will first obtain approval to approach the patient from the treating physician. Once approval is received, a co-investigator will approach them over the phone to inform the patient about a study he or she is eligible for or approach them in person during their visit. All patient eligibility data will be kept in a secure file that is password protected and secured on the Cooper secure network, in a drive behind a firewall. Only study personnel will have access to this information and the documents.

There will be four visits involved in this study, all of which follow the standard of care visit schedule:

Visit 1 is the consenting visit & patients will be consented by the study doctors or co-investigators in the clinic. The preoperative pain threshold score will be obtained.

Visit 2 is the surgery visit the patient will undergo all typical procedures as if they were not in the study. Algometer pain scores and all questionnaires (Demographics, The Tobacco, Alcohol, Prescription medications, and other Substance [TAPS] 1, Visual Analogue Scale [VAS], The 12-item Short Form Survey[SF-12], The Single Assessment Numeric Evaluation [SANE] ) must be completed by this time, either in person at Visit 1, over the phone, via REDCap , or by email prior to this visit, or in pre-op holding where they will sign official consents. The opioid consumption journal will be given to the patient for the patient to record his or her daily opioid intake immediately following TSA. The study team will ask the patients to record their daily opioid consumption in the journal for the first two weeks. Prior to prescribing any prescription narcotics post-operatively, per standard of care, The study team will utilize the Prescription Monitoring Program (PMP) to determine what prescription narcotics the patient is currently on. With the patient's permission, and on the consent form, The study team will check the patient's PMP at 3 months to record opioid consumption.

Visit 3 is the 2-week follow-up visit post-surgery. The subject's standard of care data points will be obtained at this visit, in addition to the VAS, SF-12, and SANE, again which are strictly for research purposes.

Visit 4 is the 6-week follow-up visit post-surgery. The subject would have this visit even if they were not in the study and the same procedures will be conducted during the visit as standard of care. The subject's standard of care data points will be obtained at this visit, in addition to the VAS, SF-12, and SANE, again which are strictly for research purposes.

Visit 5 is the 3-month follow-up visit post-surgery. The subject would have this visit even if they were not in the study and the same procedures will be conducted during the visit as standard of care. The subject's standard of care data points will be obtained at this visit, in addition to the VAS, SF-12, SANE, and Satisfaction Survey again which is strictly for research purposes. The hard copies of the opioid consumption journal will be collected at the final visit. The study team will not need another algometer pain score post-operative as it has already been established in the pre-operative scores.

The study team will rely on the completion of the questionnaires, opioid consumption journal, and surveys to establish a correlation between pre-operative pain threshold and postoperative outcomes. All Protected Health Information (PHI) will be kept on a secure coded document that is password encrypted and stored on the secure Cooper secure network, in a drive behind a firewall. The rest of the study-specific data will be kept on REDCap, where each patient will have a specific study identifier (ID) that corresponds with their research records. there will be no PHI stored on REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Patients who are scheduled to undergo a Total Shoulder Arthroplasty

Exclusion Criteria:

* Patients younger than 18 years
* Patients who are scheduled to undergo a Total Shoulder Arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, non-randomized observational study. There will only be one group, the treatment group, consisting of patients undergoing Total Shoulder Arthroplasty (TSA). We will recruit patients using a screen for patients who meet inclusion criteria in EPIC or recruit patients via physician referral. Inclusion criteria includes all patients over 18 years of age who are undergoing TSA. When an eligible patient is selected, we will first obtain approval to approach from the treating physician. Once approval is received, a co-investigator will approach them over the phone to inform the patient about a study he or she is eligible for or approach them in-person during their visit.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 3 months
  compare preoperative pain threshold with postoperative opioid consumption. The pain threshold will be determined using the pressure algometer/dolorimeter. The term "pain threshold" refers to the measurement of the intensity of a physical stimulus that evokes pain. To estimate the pain threshold, physical force using a mechanical stimulus will be applied with increasing intensity until the patient under evaluation refers to a pain sensation. When the patient declares that the pain is too uncomfortable, the algometer will be removed. This device will quantify the amount of force in pounds that the patient can tolerate. This number is designated as the patient's pain threshold. This value will be correlated with opioid consumption, both by self-reporting and by accessing the Prescription Monitoring Program (PMP). Opioid consumption will be quantified using milligrams of morphine equivalents (MME).
Postoperative satisfaction | 3 months
  compare preoperative pain threshold with postoperative satisfaction. The pain threshold will be determined using the pressure algometer/dolorimeter. The term "pain threshold" refers to the measurement of the intensity of a physical stimulus that evokes pain. To estimate the pain threshold, physical force using a mechanical stimulus will be applied with increasing intensity until the patient under evaluation refers to a pain sensation. When the patient declares that the pain is too uncomfortable, the algometer will be removed. This device will quantify the amount of force in pounds that the patient can tolerate. This number is designated as the patient's pain threshold. This value will be correlated with patient satisfaction. Patients will be asked how satisfied they are with their pain control. They can answer on a 1-4 scale, with 1 being the lowest satisfaction and 4 being the highest degree of satisfaction.
Postoperative return to work | 3 months
  compare preoperative pain threshold with postoperative return to work time in days.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Fedorka, MD, Principal Investigator — Cooper University Hospital Department of Orthopedics
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang MMH, Hartley RL, Leung AA, Ronksley PE, Jette N, Casha S, Riva-Cambrin J. Preoperative predictors of poor acute postoperative pain control: a systematic review and meta-analysis. BMJ Open. 2019 Apr 1;9(4):e025091. doi: 10.1136/bmjopen-2018-025091. PMID 30940757
- [Background] Friedman RJ, Eichinger J, Schoch B, Wright T, Zuckerman J, Flurin PH, Bolch C, Roche C. Preoperative parameters that predict postoperative patient-reported outcome measures and range of motion with anatomic and reverse total shoulder arthroplasty. JSES Open Access. 2019 Nov 18;3(4):266-272. doi: 10.1016/j.jses.2019.09.010. eCollection 2019 Dec. PMID 31891024
- [Background] Kim MS, Koh IJ, Sung YG, Park DC, Yoon EJ, In Y. Influence of increased pain sensitivity on patient-reported outcomes following total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2022 Mar;30(3):782-790. doi: 10.1007/s00167-021-06455-5. Epub 2021 Jan 24. PMID 33486560
- [Background] Palanisami DR, Reddy DA, Huggi V, Rajasekaran RB, Natesan R, Shanmuganathan R. Assessing Preoperative Pain Sensitivity Predicts the Postoperative Analgesic Requirement and Recovery after Total Knee Arthroplasty: A Prospective Study of 178 Patients. J Arthroplasty. 2020 Dec;35(12):3545-3553. doi: 10.1016/j.arth.2020.07.029. Epub 2020 Jul 18. PMID 32773269
- [Background] Nickel BT, Klement MR, Byrd WA, Attarian DE, Seyler TM, Wellman SS. The James A. Rand Young Investigator's Award: Battling the Opioid Epidemic with Prospective Pain Threshold Measurement. J Arthroplasty. 2018 Jul;33(7S):S3-S7. doi: 10.1016/j.arth.2018.02.060. Epub 2018 Feb 21. PMID 29567001
- [Background] Shigematsu-Locatelli M, Kawano T, Kitamura S, Nishigaki A, Yamanaka D, Aoyama B, Tateiwa H, Yokoyama M. Does preoperative patient's estimated acceptable pain affect the satisfaction with postoperative pain management? JA Clin Rep. 2017;3(1):5. doi: 10.1186/s40981-016-0075-0. Epub 2017 Jan 10. PMID 29492444
- [Background] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Background] Buchanan HM, Midgley JA. Evaluation of pain threshold using a simple pressure algometer. Clin Rheumatol. 1987 Dec;6(4):510-7. doi: 10.1007/BF02330587. PMID 3449302
- [Background] Chesterton LS, Sim J, Wright CC, Foster NE. Interrater reliability of algometry in measuring pressure pain thresholds in healthy humans, using multiple raters. Clin J Pain. 2007 Nov-Dec;23(9):760-6. doi: 10.1097/AJP.0b013e318154b6ae. PMID 18075402
- [Background] Hinarejos P, Goicoechea N, Gidi M, Leal-Blanquet J, Torres-Claramunt R, Sanchez-Soler J, Monllau JC. Pressure algometry is a suitable tool to assess anterior knee pain in osteoarthritic patients. Eur J Orthop Surg Traumatol. 2019 Jul;29(5):1089-1093. doi: 10.1007/s00590-019-02391-w. Epub 2019 Feb 7. PMID 30734099
- [Background] Sayed-Noor AS, Englund E, Wretenberg P, Sjoden GO. Pressure-pain threshold algometric measurement in patients with greater trochanteric pain after total hip arthroplasty. Clin J Pain. 2008 Mar-Apr;24(3):232-6. doi: 10.1097/AJP.0b013e3181602159. PMID 18287829